CLINICAL TRIAL: NCT01755494
Title: A Single-centre, Randomized, Open-label, Two-period, Cross-over, Bioequivalence Study of the Fixed Dose Combinations of Saxagliptin/Metformin XR Relative to Co-Administration of the Individual Components in Two Cohorts of Healthy Chinese Subjects Under Fed Conditions
Brief Title: A Bioequivalence Study of the Fixed Dose Combinations of Saxagliptin/Metformin XR Relative to Co-Administration
Acronym: SAXA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1681C00001
Record Dates: First submitted 2012-12-12; First posted 2012-12-24 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus(T2DM)
Keywords: Type 2 diabetes, Saxagliptin, Metformin,Fixed dose combination tablet, Bioequivalence, pharmacokinetic, safety, tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

ARMS (2):
- Lower dose (Experimental): co-administration of a single oral dose of a 5 mg saxagliptin tablet and a 500 mg metformin XR (Glucophage XR®) tablet vs. single FDC tablet consisting of 5 mg saxagliptin and 500 mg metformin XR (Kombiglyze XR)
  Interventions: Drug: Saxagliptin 5 mg; Drug: Metformin XR 500 mg; Drug: Komboglyze XR 5/500 mg
- Higher dose (Experimental): co-administration of a single oral dose of a 5 mg saxagliptin tablet and two (2) 500 mg metformin XR (Glucophage XR®) tablets vs. Single FDC tablet consisting of 5 mg saxagliptin and 1000 mg metformin XR (Kombiglyze XR)
  Interventions: Drug: Saxagliptin 5 mg; Drug: Mertformin XR 2 x 500 mg; Drug: Komboglyze XR 5/1000 mg

INTERVENTIONS:
Drug: Saxagliptin 5 mg — Saxagliptin oral tablet 5mg, single dose
Drug: Metformin XR 500 mg — Metformin XR oral tablet 500 mg, single dose
  Arms: Lower dose
Drug: Mertformin XR 2 x 500 mg — Metformin XR oral tablet 2 x 500 mg, single dose
  Arms: Higher dose
Drug: Komboglyze XR 5/500 mg — oral FDC tablet (saxagliptin 5 mg and metformin 500 mg), single dose
  Arms: Lower dose
Drug: Komboglyze XR 5/1000 mg — oral FDC tablet (saxagliptin 5 mg and metformin 1000 mg), single dose
  Arms: Higher dose

SUMMARY:
The primary objective of this study is to assess the pharmacokinetic parameters of saxagliptin and metformin in healthy male Chinese subjects.

DETAILED DESCRIPTION:
A Single-centre, Randomized, Open-label, Two-period, Cross-over, Bioequivalence Study of the Fixed Dose Combinations of Saxagliptin/Metformin XR Relative to Co-Administration of the Individual Components in two cohorts of Healthy Chinese Subjects under Fed Conditions

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity which is defined as having both parents and 4 grandparents who are Chinese
* Healthy male subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
* Men, ages 18 to 40 years, inclusive. The age difference among the subjects is within 10 years
* Weigh at least 50 kg and have a body mass index (BMI) between 19 and 24 kg/m2
* Sexually active fertile men must use effective birth control throughout the study and for up to 90 days after the last dose of investigational product if their partners are women of child bearing potential

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent gastrointestinal disease
* Subjects that have lymphocytopenia or thrombocytopenia
* History of autoimmune skin disorder
* Estimatedcreatinine clearance of less than 80 mL/min

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) for saxagliptin during treatment with fixed dose combination tablet of metformin plus saxagliptin compared with individual metformin XR and saxaglitpin tablets | Plasma samples at 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 hours post-dose
Maximum plasma concentration (Cmax) for metformin during treatment with fixed dose combination tablet of metformin plus saxagliptin compared with individual metformin XR and saxaglitpin tablets | Plasma samples at 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 hours post-dose
Area under plasma concentration time curve (AUC) for saxagliptin during treatment with fixed dose combination tablet of metformin plus saxagliptin compared with individual metformin XR and saxaglitpin tablets | Plasma samples at 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 hours post-dose
Area under plasma concentration time curve (AUC) for metformin during treatment with fixed dose combination tablet of metformin plus saxagliptin compared with individual metformin XR and saxaglitpin tablets | Plasma samples at 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 hours post-dose

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for 5-hydroxy saxagliptin | Plasma samples at 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 hours post-dose
Area under plasma concentration time curve (AUC) for 5-hydroxy saxagliptin | Plasma samples at 0, 15, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 and 48 hours post-dose
Safety and tolerability assessment based on medical review of AE reports:physical examination, ECG, heart rate, blood pressure, lab test | Study duration for individual subject (up to 34 days) when the safety data are collected
  Assessment for 5 mg saxagliptin co-administered with up to 1000 mg metformin XR given either separately, or as a single FDC tablet.

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Hirshberg, Study Director — Room No.: C3C-718, 1800 Concord Pike, PO Box 15437, Wilmington DE 19850-5437, USA; Haiyan Li, Principal Investigator — Peking University Third Hospital (PU3), 49 North Garden Road, Haidian District, Beijing 100191, PR. China
Locations (1):
- Research Site, Beijing, China

REFERENCES:
- See also: D1681C00001.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1189&filename=D1681C00001.pdf